CLINICAL TRIAL: NCT02465775
Title: Clinical Study to Evaluate the Performance of the UltraShape Device for Fat Reduction Treatment in the Flanks Area vs. Control
Brief Title: Fat Reduction in the Flanks Area vs. Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF18361
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Flanks Fat Reduction vs. Control
Keywords: non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UltraShape treatment in all subjects (Experimental): UltraShape treatment for fat reduction to unilateral flank for all subjects with untreated flank as control.
  Interventions: Device: UltraShape treatment

INTERVENTIONS:
Device: UltraShape treatment — Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time.
  Other Names: Contour V1

SUMMARY:
Prospective, blinded, one arm, baseline-controlled clinical study for the evaluation the performance of the UltraShape treatment for non-invasive fat reduction by compare control and treated flanks.

Study subjects will undergo UltraShape treatments on one randomized flank using the U-Sculpt/VDF Transducer. The second flank will not be treated (control). Both flanks (treated and control) will be compared to baseline, as well as, one to each other

DETAILED DESCRIPTION:
This study is a prospective, baseline and blinded controlled, comparison, clinical study showing the performance and safety of the UltraShape treatment for non-invasive fat reduction at the flanks area comparing improvement observed in treated versus control flanks.

Up to 60 Healthy subjects in up to 4 investigational sites will be enrolled in this study. All subjects will undergo an assessment of their general health. During the treatment period, subject's fat thickness will be measured on both flanks. Three successive bi-weekly (two weeks interval) UltraShape treatments will be performed on one randomized flank, while the second flank will not be treated and served as a control.

The study subjects will undergo UltraShape treatments on one flank using the U-Sculpt /VDF Transducer, the treated flank will remain steady along the study and will be comparing to the baseline and to the controlled flank Three follow-up visits will be conducted as follows: 4 weeks (4wk FU), 8 weeks (8wk FU) and 16 weeks (16wk FU) post last treatment (Tx.3).

Subject's fat thickness will be measured on both flanks in the measurements points using caliper at each visit (at treatment visits, prior to treatment). Ultrasound measurements will be taken at each visit, except for the second treatment visit, on each flank. Investigator satisfaction will be assessed at all FU visits. In addition, subject questionnaires will be completed at each follow-up visit. Photographs of the front, right, left and back view of each flank will be performed under visible light conditions at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, between 18 to 60 years of age at the time of enrolment
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
5. BMI interval: BMI between 22 to 30 (normal to overweight, but not obese).
6. If female, not pregnant or lactating, must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative urine pregnancy test as tested before each treatment and at the last follow-up visit for women with child-bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
11. Very poor skin quality (i.e., severe laxity)
12. Abdominal wall diastasis or hernia on physical examination
13. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
14. Obesity (BMI above 30)
15. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
17. Fat thickness lower than 2.5 cm after strapping at the treated area.
18. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trial/s).
19. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of flank fat reduction vs. control | up to 16 weeks after treatment
  Evaluate the efficacy of UltraShape treatments with the U-sculpt/VDF Transducer for flanks fat reduction as assessed by comparing the change during the study on the treated flank area and compare to the change observed on the un-treated (control) flank

SECONDARY OUTCOMES:
Fat thickness reduction on the treated flank | 4, 8 and 16 weeks
  measured by caliper and by Ultrasound device
Investigator satisfaction assessment | 4, 8 and 16 weeks
  5-Point Likert Scale
Subject satisfaction assessment | 4, 8 and 16 weeks
  Subjects will answer the questionnaire
pain assessment | day 0, 2 weeks and 4 weeks
  NSR scale
Safety of flank fat reduction | up to 20 weeks after treatment
  Evaluate the safety of the treatment with the UltraShape device using the U-Sculpt/VDF Transducer for flanks treatment area

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weiss, MD, Principal Investigator — 54 Scot Adams Road, Hunt Valley Baltimore USA; William P. Colem, MD, Principal Investigator — Coleman Center for Cosmetic Dermatologic Surgery
Locations (3):
- United States (3):
  - Coleman Center for Cosmetic Dermatologic Surgery, Metairie, Louisiana
  - Maryland Laser, Skin, & Vein Institute, LLC, Hunt Valley, Maryland
  - Gold Skincare, Nashville, Tennessee

REFERENCES:
- [Background] Arner P. Regional adipocity in man. J Endocrinol. 1997 Nov;155(2):191-2. doi: 10.1677/joe.0.1550191. No abstract available. PMID 9415044
- [Background] Gasparotti M. Superficial liposuction: a new application of the technique for aged and flaccid skin. Aesthetic Plast Surg. 1992 Spring;16(2):141-53. doi: 10.1007/BF00450606. PMID 1570777